CLINICAL TRIAL: NCT04083755
Title: Impact of Intravenous Iron Treatment of Preoperative Anemia in Patients With Lower Extremity Peripheral Artery Disease
Brief Title: Impact of Intravenous Iron Treatment of Preoperative Anemia in Patients With LEAD (IRONPAD)
Acronym: IRONPAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biobizkaia Health Research Institute (Other Government)
Collaborators: Sociedad Espanola de Angiologia y Cirugia Vascular (Network)
Responsible Party: Principal Investigator, Ana Apodaka Diez, Vascular Surgeon, Biobizkaia Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-003714-40; 2018-003714-40 (EudraCT Number)
Record Dates: First submitted 2019-09-01; First posted 2019-09-10 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Anemia; Peripheral Arterial Occlusive Disease
Keywords: anemia; iron; surgery; PAD
MeSH Terms: conditions — Anemia; Peripheral Arterial Occlusive Disease 1 | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Line A (Active Comparator): One dose of Ferric carboxymaltose (1000mg) intravenous. Duration of administration 15 minutes.
  Interventions: Drug: Ferric Carboxymaltose Injection [Injectafer]
- Line B (Other): No treatment or treatment oral with iron supplementation if iron-deficiency anemia
  Interventions: Other: no treatment or oral iron supplementation

INTERVENTIONS:
Drug: Ferric Carboxymaltose Injection [Injectafer] — 1000mg intravenous
  Other Names: Ferinject
  Arms: Line A
Other: no treatment or oral iron supplementation — No treatment or treatment oral with iron supplementation if iron-deficiency anemia
  Arms: Line B

SUMMARY:
Introduction: Anaemia due to iron and vitamin deficiency among patients with critical limb ischemia is high (>50%). The prevalence of a higher rate of anaemia extends into the three months prior to revascularization surgery, it is associated with longer hospital stays and more transfusions in addition to being a factor in poor prognoses. Study and treatment of anaemia within the perioperative period could improve the surgical outcomes, including the recovery and the quality of patients' lives. There are several types of intravenous iron preparations with different administration protocols, but there is not a consensus on the timing and type of the appropriate iron therapy. To the best of our knowledge, there is no data on the performance of intravenous iron in the management of preoperative anaemia in patients with peripheral artery disease (PAD) in vascular surgery.

Methods and analysis: The IRONPAD Study is a phase IV randomised controlled trial with two branches of treatment on the efficacy of intravenous iron therapy for the optimisation of blood use and prognosis in the perioperative period of patients with anaemia undergoing revascularisation for chronic lower limb ischemia. The study randomises 240 patients with anaemia to: treat with a single intravenous dose of ferric carboxymaltose (1000 mg) or no treatment vs oral iron supplements (if severe anaemia) a minimum of two days prior to lower limb revascularisation surgery. The primary outcome is to reduce the incidence of transfusion from randomisation up to 30+7 days after the main surgery. The secondary outcomes will be included to establish the optimal preoperative moment of increased intravenous iron administration, to raise haemoglobin levels; to study the evolution of haemoglobin from inclusion to 30+7 days after surgery; and to determine the impact of anaemia and its treatment on the length of hospital stay, morbidity and mortality, as well as the quality of life in this period.

DETAILED DESCRIPTION:
The IRONPAD Study is a phase IV randomised controlled trial with two branches of treatment on the efficacy of intravenous iron therapy for the optimisation of blood use and prognosis in the perioperative period of patients with anaemia undergoing revascularisation for chronic lower limb ischemia.

Patients admitted to hospital with anaemia and indication of elective revascularisation surgery for chronic ischemia of the lower limbs will be eligible for screening. Anaemia in this study is established following the WHO criteria with haemoglobin (Hb) <130 g/L in men and <120 g/L in women 21.

Patients will be selected according to the usual practice, without excluding patients because of comorbidity or other reasons that may affect results (selection bias).

Prior to inclusion, freely given written informed consent will be obtained from all patients. Once included, each patient will be masked into a unique identity number (correlative according to inclusion), as a reference of patient ID in the registry.

Each patient will be randomised to a line A or line B of treatment.

* Line A: a single, ferric carboxymaltose (Ferinject®) 1000 mg IV iron dose administration. The infusion will be according to product specifications with an approximate duration of 15 minutes during hospitalisation and will not require an additional site visit or extended period of hospitalisation.
* Line B: control. The control group will not receive specific treatment. In case of severe iron deficiency anaemia, oral iron supplements (iron sulphate dihydrate) will be given.

Both lines may be followed in addition to taking vitamin B12 and folic acid, if indicated.

The patient, once included in the study, may receive a blood transfusion if the following criteria are met:

- Absolute indication: Hemodynamic instability Active bleeding Hb <7 g/dl

- Relative indications: in case of Hb <8.5 g/dL or haematocrit <28% following the clinical criteria of the medical specialist.

Interventions to be measured:

The data collected at baseline will include patients' past medical history, medications, blood tests (including hemogram, iron tests and renal function), comorbidity index (Charlson Scale), lower limbs chronic ischemia category and the limb scheduled for revascularisation (including registry of any trophic lesions and if they have signs of active infection), height, weight and body-mass index of the patient. In addition, already validated quality of life questionnaire, the Short Form-36 Health Survey (SF-36) will be completed.

Procedure data will record: date of IV iron treatment, if received, dose and any adverse events during or after administration; ASA (American Society of Anaesthesiologists) risk level; type of surgery performed for revascularisation of lower limbs, information on clinical success and complications of the intervention. Blood records will include haemoglobin before and first day after surgery and number of red blood cell units of or any other blood component transfused during the surgical procedure. If surgery does not finally take place, data from the 30 days after inclusion will be registered for analysis with intention to treat.

The hospital discharge visit will record: date of discharge; last hemogram; number of blood transfusions from the postoperative period until discharge; days in intensive care; adverse events such as medical and surgical complications as well as mortality.

The final follow-up visit will take place 30 days after the main surgery (with + 7 day window) it would be performed by telephone, in the outpatient consultation or in the hospital if the patient continues to be hospitalised; in that case, the discharge visit and final visit will be made simultaneously. It will record: blood tests (including hemogram, iron tests), clinical success, serious adverse events (SAE) and mortality, which may have occurred between hospital discharge and the visit in addition to Short Form-36 Health Survey (SF-36). See Fig. 1 for Assessment flow diagram.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes over 18 years
* Patients diagnosed with anemia, considered as Hb <13.0 g/dL in mens and Hb<12g/dL in women
* Patients diagnosed with symptomatic chronic lower limb ischemia (degrees 2-5 by Rutherford-Baker, both included, Fontaine II-IV), who will undergo surgical revascularization (endovascular or open) and accept treatment
* Revascularization surgery scheduled in the approximate minimum period of two days, (> 48 hours) from the inclusion, Patients diagnosed with iron deficiency anemia being treated with oral iron in their usual medication and with inadequate iron storage for surgical intervention (ferritin <100 ng/ml) or functional iron deficiency: ferritin 100-500 ng/ml with TSI < 20% .
* They are able and willing to give written informed consent at the time of selection

Exclusion Criteria:

* Patients with acute ischemia will be excluded
* Severe anemia < 8 gr/dL
* Arterial hypertension not controlled with antihypertensive medication (considered with systolic blood pressure> 180mmHg or diastolic> 100mmHg)
* Acute renal failure or renal failure with creatinine clearance <30mmHg
* Patient with documented intolerance or allergy to iron or its derivatives
* Unstable angina, defined as electrocardiographic changes with chest pain that indicate resting myocardial ischemia
* History of stroke in the previous 6 months
* Patients with thrombocytopenia less than 50,000ug/dl or alterations in coagulation
* That you are simultaneously participating in a clinical trial that conditions or modifies the registry
* Pregnancy or lactation (pregnancy tests in women of childbearing age according to usual practice)
* Rejection of treatment or inclusion in the registry by the patient
* Patients who refuse to receive transfusions of blood products (for example, Jehovah's Witnesses)
* Patients with criteria of SEPSIS
* Patients with Ferritin <30 ng/ml that will be directed for digestive study
* Patients with active neoplasia
* Probable or confirmed case with active SARS-CoV-2 infection
* Patients who are not able to give their informed consent or understand the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To reduce the incidence of transfusion (receiving any volume of 1 unit or more than 1 unit of packed red cells) from randomisation up to 30 days (with +/- 15-day window) after the main surgery | From inclusion date to 30 days (with +7 window) after the main surgery
  Number of red blood cell units of or any other blood component transfused during the surgical procedure and from the postoperative period until discharge. If surgery does not finally take place, data from the 30 days after inclusion will be registered for analysis with intention to treat.

SECONDARY OUTCOMES:
Changes and evolution of hemoglobin during admission; difference in hemoglobin (Hb) between inclusion, intervention and discharge. | From inclusion date to 30 days (with +7day window) after surgical procedure
  The data collected at baseline will include patients blood tests (including hemogram). Blood records during surgical period will include haemoglobin (g/dL) before and first day after surgery. (If surgery does not finally take place, data from the 30 days after inclusion will be registered for analysis with intention to treat).The final follow-up visit will take place 30 days after the main surgery it would be performed by telephone, in the outpatient consultation or in the hospital if the patient continues to be hospitalised; in that case, the discharge visit and final visit will be made simultaneously. It will record: blood tests (including hemogram).
Establish the optimal preoperative moment of increased intravenous iron yield to increase Hb | From inclusion date to 30 days (with +7 window) after the main surgery
  Best time before surgery for treatment anemia with ferric carboxymaltose
Impact of anemia and its treatment on the length of hospital stay | From inclusion date to 30 days (with +7 window) after the main surgery
  Difference between both groups in days of hospitalization after main surgery
Impact of anemia and its treatment on morbidity | From inclusion date to 30 days (with +7 window) after the main surgery
  Serious adverse events such, as medical and surgical complications during hospitalization and at final follow-up visit (which may have occurred between hospital discharge and final the visit).
Impact of anemia and its treatment on mortality | From inclusion date to 30 days (with +7 window) after the main surgery
  Death and cause, if known, during hospitalization and at the final follow-up visit (which may have occurred between hospital discharge and final the visit).
Impact of anemia and its treatment on quality of life | From inclusion date to 30 days (with +7 window) after the main surgery
  The Short Form-36 Health Survey (SF-36) will be completed at inclusion and at the final visit that will take place 30 days after the main surgery (with +/- 15-day window). It would be performed by telephone, in the outpatient consultation or in the hospital if the patient continues to be hospitalized.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Apodaka Diez, MD, Principal Investigator — Vascular Surgeon; Jose Manuel Rodriguez Chinesta, MD, Principal Investigator — Internal Medicine
Locations (5):
- Spain (5):
  - Hospital de Galdakao-Usansolo., Galdakao, Basque Country
  - Servicio de Angiología y Cirugía vascular del Hospital Universitario Cruces, Barakaldo, Biscay
  - Hospital de Getafe, Getafe, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be send to publication in the next months
Supporting Information: Study Protocol
Time Frame: open access to read as soon as published
Access Criteria: open

REFERENCES:
- [Background] Esteban Gracia C, Escudero Rodríguez JR, Preciado Mora MJ, et al. Prevalencia de anemia en pacientes sometidos a cirugía vascular electiva y su influencia en el postoperatorio. Angiologia 2016;68:396-404. doi:10.1016/j.angio.2016.01.015
- [Background] Vega de Ceniga M, Bravo E, Izagirre M, Casco C, Estallo L, Esteban M, Barba A. Anaemia, iron and vitamin deficits in patients with peripheral arterial disease. Eur J Vasc Endovasc Surg. 2011 Jun;41(6):828-30. doi: 10.1016/j.ejvs.2011.01.017. Epub 2011 Feb 25. PMID 21353606
- [Background] Gonzalez ZM, Barrasa AG, Renau AR. [Anaemia, iron, transfusion and therapeutic alternatives. A review from a surgical perspective]. Cir Esp. 2010 Dec;88(6):358-68. doi: 10.1016/j.ciresp.2010.03.014. Epub 2010 May 11. Spanish. PMID 20462573
- [Background] Musallam KM, Tamim HM, Richards T, Spahn DR, Rosendaal FR, Habbal A, Khreiss M, Dahdaleh FS, Khavandi K, Sfeir PM, Soweid A, Hoballah JJ, Taher AT, Jamali FR. Preoperative anaemia and postoperative outcomes in non-cardiac surgery: a retrospective cohort study. Lancet. 2011 Oct 15;378(9800):1396-407. doi: 10.1016/S0140-6736(11)61381-0. Epub 2011 Oct 5. PMID 21982521
- [Background] Munoz M, Gomez-Ramirez S, Martin-Montanez E, Pavia J, Cuenca J, Garcia-Erce JA. Perioperative intravenous iron: an upfront therapy for treating anaemia and reducing transfusion requirements. Nutr Hosp. 2012 Nov-Dec;27(6):1817-36. doi: 10.3305/nh.2012.27.6.6087. PMID 23588429
- [Background] Baron DM, Hochrieser H, Posch M, Metnitz B, Rhodes A, Moreno RP, Pearse RM, Metnitz P; European Surgical Outcomes Study (EuSOS) group for Trials Groups of European Society of Intensive Care Medicine; European Society of Anaesthesiology. Preoperative anaemia is associated with poor clinical outcome in non-cardiac surgery patients. Br J Anaesth. 2014 Sep;113(3):416-23. doi: 10.1093/bja/aeu098. Epub 2014 May 14. PMID 24829444
- [Background] Fowler AJ, Ahmad T, Phull MK, Allard S, Gillies MA, Pearse RM. Meta-analysis of the association between preoperative anaemia and mortality after surgery. Br J Surg. 2015 Oct;102(11):1314-24. doi: 10.1002/bjs.9861. PMID 26349842
- [Background] Glance LG, Dick AW, Mukamel DB, Fleming FJ, Zollo RA, Wissler R, Salloum R, Meredith UW, Osler TM. Association between intraoperative blood transfusion and mortality and morbidity in patients undergoing noncardiac surgery. Anesthesiology. 2011 Feb;114(2):283-92. doi: 10.1097/ALN.0b013e3182054d06. PMID 21239971
- [Background] Zollo RA, Eaton MP, Karcz M, Pasternak R, Glance LG. Blood transfusion in the perioperative period. Best Pract Res Clin Anaesthesiol. 2012 Dec;26(4):475-84. doi: 10.1016/j.bpa.2012.10.001. PMID 23351234
- [Background] Kougias P, Orcutt S, Pak T, Pisimisis G, Barshes NR, Lin PH, Bechara CF. Impact of postoperative nadir hemoglobin and blood transfusion on outcomes after operations for atherosclerotic vascular disease. J Vasc Surg. 2013 May;57(5):1331-7; discussion. doi: 10.1016/j.jvs.2012.10.108. Epub 2013 Feb 4. PMID 23384496
- [Background] Dunkelgrun M, Hoeks SE, Welten GM, Vidakovic R, Winkel TA, Schouten O, van Domburg RT, Bax JJ, Kuijper R, Chonchol M, Verhagen HJ, Poldermans D. Anemia as an independent predictor of perioperative and long-term cardiovascular outcome in patients scheduled for elective vascular surgery. Am J Cardiol. 2008 Apr 15;101(8):1196-200. doi: 10.1016/j.amjcard.2007.11.072. Epub 2008 Feb 7. PMID 18394458
- [Background] Desormais I, Aboyans V, Bura A, Constans J, Cambou JP, Messas E, Labrunie A, Lacroix P. Anemia, an independent predictive factor for amputation and mortality in patients hospitalized for peripheral artery disease. Eur J Vasc Endovasc Surg. 2014 Aug;48(2):202-7. doi: 10.1016/j.ejvs.2014.04.005. Epub 2014 Jun 14. PMID 24935912
- [Background] Toor IS, Jaumdally RJ, Moss MS, Babu SB. Preprocedural hemoglobin predicts outcome in peripheral vascular disease patients undergoing percutaneous transluminal angioplasty. J Vasc Surg. 2009 Aug;50(2):317-21. doi: 10.1016/j.jvs.2009.03.041. PMID 19631867
- [Background] Preciado Mora MJ, Azparren Cabezón G, Escudero Rodríguez JR, et al. La anemia como factor de riesgo quirúrgico en cirugía vascular. Algoritmos de diagnóstico y tratamiento. Angiologia 2017;69:242-9. doi:10.1016/j.angio.2016.08.007
- [Background] Kumar A. Perioperative management of anemia: limits of blood transfusion and alternatives to it. Cleve Clin J Med. 2009 Nov;76 Suppl 4:S112-8. doi: 10.3949/ccjm.76.s4.18. PMID 19880828
- [Background] Cuenca J, Garcia-Erce JA, Martinez AA, Solano VM, Molina J, Munoz M. Role of parenteral iron in the management of anaemia in the elderly patient undergoing displaced subcapital hip fracture repair: preliminary data. Arch Orthop Trauma Surg. 2005 Jun;125(5):342-7. doi: 10.1007/s00402-005-0809-3. Epub 2005 Mar 24. PMID 15789233
- [Background] Serrano-Trenas JA, Ugalde PF, Cabello LM, Chofles LC, Lazaro PS, Benitez PC. Role of perioperative intravenous iron therapy in elderly hip fracture patients: a single-center randomized controlled trial. Transfusion. 2011 Jan;51(1):97-104. doi: 10.1111/j.1537-2995.2010.02769.x. PMID 20630042
- [Background] Froessler B, Palm P, Weber I, Hodyl NA, Singh R, Murphy EM. The Important Role for Intravenous Iron in Perioperative Patient Blood Management in Major Abdominal Surgery: A Randomized Controlled Trial. Ann Surg. 2016 Jul;264(1):41-6. doi: 10.1097/SLA.0000000000001646. PMID 26817624
- [Background] Hallet J, Hanif A, Callum J, Pronina I, Wallace D, Yohanathan L, McLeod R, Coburn N. The impact of perioperative iron on the use of red blood cell transfusions in gastrointestinal surgery: a systematic review and meta-analysis. Transfus Med Rev. 2014 Oct;28(4):205-11. doi: 10.1016/j.tmrv.2014.05.004. Epub 2014 Jun 3. PMID 24997001
- [Background] Ng O, Keeler BD, Mishra A, Simpson A, Neal K, Brookes MJ, Acheson AG. Iron therapy for pre-operative anaemia. Cochrane Database Syst Rev. 2015 Dec 22;(12):CD011588. doi: 10.1002/14651858.CD011588.pub2. PMID 26694949
- [Background] Nutritional anaemias. Report of a WHO scientific group. World Health Organ Tech Rep Ser. 1968;405:5-37. No abstract available. PMID 4975372
- [Background] Esteban C, Rodriguez P, Escudero JR, Clara A, Fernandez A, Fernandez S, Agundez I. Anaemia in patients who underwent vascular surgery: a significant predictor of amputation and death. Med Clin (Barc). 2019 Jan 4;152(1):6-12. doi: 10.1016/j.medcli.2018.01.029. Epub 2018 Apr 9. English, Spanish. PMID 29650265
- [Background] Munoz M, Gomez-Ramirez S, Besser M, Pavia J, Gomollon F, Liumbruno GM, Bhandari S, Cladellas M, Shander A, Auerbach M. Current misconceptions in diagnosis and management of iron deficiency. Blood Transfus. 2017 Sep;15(5):422-437. doi: 10.2450/2017.0113-17. PMID 28880842
- [Background] Dignass AU, Gasche C, Bettenworth D, Birgegard G, Danese S, Gisbert JP, Gomollon F, Iqbal T, Katsanos K, Koutroubakis I, Magro F, Savoye G, Stein J, Vavricka S; European Crohn's and Colitis Organisation [ECCO]. European consensus on the diagnosis and management of iron deficiency and anaemia in inflammatory bowel diseases. J Crohns Colitis. 2015 Mar;9(3):211-22. doi: 10.1093/ecco-jcc/jju009. Epub 2014 Dec 3. No abstract available. PMID 25518052
- [Background] Goodnough LT, Shander A, Spivak JL, Waters JH, Friedman AJ, Carson JL, Keating EM, Maddox T, Spence R. Detection, evaluation, and management of anemia in the elective surgical patient. Anesth Analg. 2005 Dec;101(6):1858-1861. doi: 10.1213/01.ANE.0000184124.29397.EB. PMID 16301274
- [Background] Kotze A, Harris A, Baker C, Iqbal T, Lavies N, Richards T, Ryan K, Taylor C, Thomas D. British Committee for Standards in Haematology Guidelines on the Identification and Management of Pre-Operative Anaemia. Br J Haematol. 2015 Nov;171(3):322-31. doi: 10.1111/bjh.13623. Epub 2015 Sep 6. No abstract available. PMID 26343392
- [Background] Edwards TJ, Noble EJ, Durran A, Mellor N, Hosie KB. Randomized clinical trial of preoperative intravenous iron sucrose to reduce blood transfusion in anaemic patients after colorectal cancer surgery. Br J Surg. 2009 Oct;96(10):1122-8. doi: 10.1002/bjs.6688. PMID 19731228
- [Background] Kim YH, Chung HH, Kang SB, Kim SC, Kim YT. Safety and usefulness of intravenous iron sucrose in the management of preoperative anemia in patients with menorrhagia: a phase IV, open-label, prospective, randomized study. Acta Haematol. 2009;121(1):37-41. doi: 10.1159/000210062. Epub 2009 Mar 31. PMID 19332985
- [Background] Rognoni C, Venturini S, Meregaglia M, Marmifero M, Tarricone R. Efficacy and Safety of Ferric Carboxymaltose and Other Formulations in Iron-Deficient Patients: A Systematic Review and Network Meta-analysis of Randomised Controlled Trials. Clin Drug Investig. 2016 Mar;36(3):177-94. doi: 10.1007/s40261-015-0361-z. PMID 26692005
- [Background] Friedrisch JR, Cancado RD. Intravenous ferric carboxymaltose for the treatment of iron deficiency anemia. Rev Bras Hematol Hemoter. 2015 Nov-Dec;37(6):400-5. doi: 10.1016/j.bjhh.2015.08.012. Epub 2015 Oct 14. PMID 26670403